CLINICAL TRIAL: NCT04995770
Title: Text Messages for Adolescent and Young Adult Liver Transplant Recipients
Brief Title: Text Messages for Liver Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Caitlin Sayegh, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHLA-19-00189
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Medication Adherence; Liver Transplant Disorder
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider
Masking Description: Transplant coordinators were masked from intervention assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Praise Text Messages (Experimental): The text message praise intervention lasted for 6 months. Each week, transplant coordinators, masked from who enrolled in the study or to which condition participants were randomized, prepared a list of all patients in the study age group whose laboratory blood tests indicated that immunosuppressant medications were within the expected range. A researcher reviewed the list to identify whether any of patients were currently assigned to the intervention, and if so, sent text message praise via REDCap's text message function. We rotated through 14 standardized text messages each week. Examples of messages included: "Your labs look very good. Super job taking your meds!" and "Your labs look great! Thanks for putting in the effort to take care of your health!."
  Interventions: Behavioral: Praise Text Messages
- Usual Care (No Intervention): Participants in the usual care arm did not receive any praise text messages. All participants continued to receive usual care from the multidisciplinary liver transplant team, including phone calls and follow-up care when laboratory blood tests indicated that immunosuppressant medications were outside of the expected range.

INTERVENTIONS:
Behavioral: Praise Text Messages — Texting messages with praise content, to positive reinforce medication adherence
  Arms: Praise Text Messages

SUMMARY:
Although medical advancements have enabled children experiencing liver transplants to live longer, medical management post-transplant is ongoing and complex. Many findings underscore adolescents as being a particularly vulnerable population, with rates of nonadherence being four times higher than in adults. This pilot study aims to explore the feasibility and impact of a brief text-messaging intervention in a randomized controlled trials (N = 50). We have three primary aims: 1) Study patient satisfaction with and utilization of this intervention in order to better understand feasibility and acceptability; 2) Investigate the effects of this intervention on medication adherence, healthcare utilization, and health status; and 3) Examine potential effects of the intervention on the physician-patient relationship, motivation for adherence, and other variables.

DETAILED DESCRIPTION:
The proposed randomized control pilot study will be based at the Liver Transplant Clinic at CHLA. Approximately 25 participants will be randomly assigned to the intervention arm, whereas 25 participants will be assigned to treatment as usual (TAU), for a total sample size of N = 50. As there are approximately 90 patients who meet inclusion criteria currently in care, recruiting 50 for this study is feasible. The intervention will last for six months. During this time, participants in the intervention arm will receive a brief text-message on their cell-phones whenever laboratory blood tests indicate that immunosuppressant medications are within the expected range. This will primarily be measured via trough levels of calcineurin inhibitors, but will also take into account complete blood count, comprehensive metabolic panel, and magnesium level results, as reviewed by the transplant physician. The purpose of these text messages is to alert participants that physicians are indeed checking participant liver levels and recognizing when participants are putting in the work to keep themselves healthy. Multiple standardized text messages will be created so that participants do not receive identical ones each time. An example text message may include "Your liver levels have been checked and look good. The effort you are putting into taking your meds shows!" Participants in the TAU arm will not receive any text messages.If trough levels or any other study measure indicates possible nonadherence, nonadherence will still be addressed by their physicians, social work, or whatever is indicated per clinic standard of care. Furthermore, additional psychosocial or medical support will not be withheld from patients whose labs indicate nonadherence for either the intervention or TAU arms.

All participants will complete questionnaires at four points: Baseline, mid-way through the intervention period (three-months), immediately after the conclusion of the intervention (six-months), and three months post-intervention. Participants will complete self-report measures assessing medication adherence (Visual Analogue Scale), participants' sense of trust in their medical providers (Trust in Physician Scale) and motivation for medication adherence (Rollnick's Readiness Ruler). In addition, participants will complete self-reported measures of anxiety (General Anxiety Disorder-7), depression (Patient Health Questionnaire-9), and socioeconomic status (Family Affluence Scale II). Several variables will also be abstracted from the electronic medical record, from one year prior to study enrollment to one year post study enrollment. At the end of the intervention, participants will complete an exit survey assessing its feasibility and acceptability. They will be asked to discuss which components of the intervention were most helpful, so this information can be used for possible dismantling study approaches in the future. Twenty-five participants will also be randomly selected and asked to participate in a 30-60 minute telephone interview in order to assess feasibility and acceptability of the study, as well as gain their insight regarding potentially helpful future interventions. Medical or psychosocial support will not be withheld from patients who drop out of the study or do not complete study measures. All data will be collected via Redcap, a HIPAA-compliant on-line platform that will allow participants to complete measures securely on-line at home.

ELIGIBILITY:
Inclusion Criteria:

* having a liver transplant
* receiving care at Children's Hospital Los Angeles
* having access to a working cellphone
* speaking English.

Exclusion Criteria:

* insufficient cognitive capacity to understand or engage in the procedures of the study

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
Self-Reported Medication Adherence | 9 months
  Visual Analogue Scale (0-100% range, with higher scores indicating better values)
Medication Variability Observed in Immunosuppressant Labs | 12 months
  medication level variability index (calculated as standard deviation of at least 3 lab values, with lower scores indicating better values)

SECONDARY OUTCOMES:
Motivation for Adherence | 9 months
  Rollnick's Readiness Ruler (0-10 range, with higher scores indicating better values)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walsh JC, Dalton M, Gazzard BG. Adherence to combination antiretroviral therapy assessed by anonymous patient self-report. AIDS. 1998 Dec 3;12(17):2361-3. No abstract available. PMID 9863888
- [Background] Rollnick S, Miller WR, Butler C. Motivational interviewing in health care: helping patients change behavior. Guilford Press; 2008.
- [Background] Shemesh E, Fine RN. Is calculating the standard deviation of tacrolimus blood levels the new gold standard for evaluating non-adherence to medications in transplant recipients? Pediatr Transplant. 2010 Dec;14(8):940-3. doi: 10.1111/j.1399-3046.2010.01396.x. Epub 2010 Oct 1. PMID 20887400